CLINICAL TRIAL: NCT06816420
Title: Effect Of Local Cold Applıcatıon On Paın and Vıtal Sıgns Durıng Port Catheter Needle Insertıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gulden Basit, Doç.Dr. Gülden BASİT, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23841101021
Record Dates: First submitted 2025-01-26; First posted 2025-02-10 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Catheter Placement and Perceived Pain; Vital Sign Monitoring; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: one group will be applied cold application, and the other group will not.
Who Masked: Outcomes Assessor
Masking Description: Study result will be analysed by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Applıcatıon (Experimental): After information about the study is provided through the informed consent form and participation approval is obtained, privacy is ensured in a single room and according to the literature review, cold application will be applied to all patients by the same nurse with ice gel for 1 minute before the application, centered on the area where the reservoir part of the port catheter is located.
  Interventions: Other: Cold Application
- control (No Intervention): There will be no cold application before port catheter needle insertion in this group.

INTERVENTIONS:
Other: Cold Application — The effects of local cold application on pain and vital signs during port catheter needle insertion will be studied in this group.
  Arms: Cold Applıcatıon

SUMMARY:
In this study, the effect of cold application on the pain experienced during port catheter needle insertion and the change in the patient's vital signs will be evaluated. It is thought that with this application, patients will experience less pain during port catheter needle insertion. The change in the patient's vital signs and pain status will also be evaluated. The research will be conducted in the outpatient chemotherapy department of a Hospital.

DETAILED DESCRIPTION:
The effects of lidocaine cream, cryotherapy (cold application to the skin), cutaneous stimulation therapy (pressure and massage) methods , virtual reality application and aromatherapy applied via inhalation on reducing pain were investigated in order to reduce the pain during port catheter needle insertion. In this study, the effect of cold application on the pain experienced during port catheter needle insertion and the change in the patient's vital signs will be evaluated. It is thought that with this application, patients will experience less pain during port catheter needle insertion. The change in the patient's vital signs according to the pain status will also be evaluated. The research will be conducted in the outpatient chemotherapy department of Necmettin Erbakan University Faculty of Medicine Hospital. The universe of the research will consist of all patients with port catheters in the outpatient chemotherapy department of Necmettin Erbakan University Faculty of Medicine Hospital. The sample of the research will consist of patients who meet the inclusion criteria and agree to participate in the research.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 18-65, who are pain-free, receiving treatment in an outpatient chemotherapy unit, who have a port catheter, who have a Huber port needle of L (large) 20 mm-20 gauge, and who can read and write in Turkish.

Exclusion Criteria:

Patients taking "oxaliplatin" Patients aged 65 and over Patients who have started using a port catheter but whose stitches have not yet healed Patients who have not passed 30 days since the port catheter was inserted Patients with any redness, swelling or tenderness in the port catheter area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Pain level | before and in ten minutes after cold application
  patients pain levels will be assessed with a Visual analogue scale (0-10 point)
Vıtal Sıgns (blood pressure, mm/Hg) | before and in ten minutes after cold application
  blood pressure will be evaluated with an electronic device
Vıtal Sıgns (body temperature, Celcius degree) | before and in ten minutes after cold application
  body temperature will be evaluated with an electronic device
Vıtal Sıgns (pulse rate in one minutes) | before and in ten minutes after cold application
  pulse rate will be evaluated by researchers manually.
vital signs (saturation rate, %) | before and in ten minutes after cold application
  saturation rate will be evaluated with using a pulse meter

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Basit, Assoc. Prof., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research data can be requested from the authors.